CLINICAL TRIAL: NCT01327157
Title: Neuro Occlusal Rehabilitation in Patient With Peripheral Facial Paralysis - a Randomized Clinical Trial
Brief Title: Study of a New Technique to Improve the Symptoms of Orofacial Discomfort in Patients With Peripheral Facial Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rosana de Queiroz, Rosana de Queiroz Costa, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 0323/08
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Peripheral Nerve Facial Nerve Paralysis; Facial Nerve Diseases; Orofacial Pain
Keywords: Facial Paralysis / rehabilitation.; Dental Occlusion.; Occlusal Adjustment.; Malocclusion / therapy.
MeSH Terms: conditions — Facial Nerve Diseases; Facial Pain; Facial Paralysis; Bites and Stings; Malocclusion | interventions — Occlusal Adjustment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visual Analog Scale (VAS) (Placebo Comparator): Initial consultation, dental cleaning and performing the visual analog scale. Consultation three months after achieving "visual analog scale" final
  * VAS and dental cleaning at the first query.
  * VAS at the last query. In the second period (91-180 days) that participants have been moved from the Placebo group (VAS) to the Experimental group(Occlusal Adjustment).
  Interventions: Behavioral: Visual analog scale.
- Occlusal adjustment (Experimental): In all consultations, was performed VAS and occlusal adjustment. Three sessions of intervention are doing. The Gnathostatic models were performed in the first and last query. To reach a terminal axis of rotation of the jaw the patient to perform the act of swallowing for 3 times, and after palpation of the muscles, masseter and temporal on both sides and compared with the marks of carbon found in the teeth and started the adjustment following the rules of Guichet with a cylindrical drill with a thin cut.. The rules to guide the occlusal adjustment selective grinding were in this sequence: Occlusal adjustment to the centric relation: with sliding towards anterior; with sliding towards the medium line; with sliding opposite to the medium line; No sliding.
  Interventions: Procedure: occlusal adjustment.; Behavioral: Visual analog scale.

INTERVENTIONS:
Procedure: occlusal adjustment. — It prompted the patient to perform the act of swallowing for 3 times to reach a terminal axis of rotation of the jaw and from this to start. Will be held palpation of the muscles, masseter and temporal on both sides and compared with the marks of carbon found in the teeth. After starts the adjustment following the rules of Guichet with a cylindrical drill with a thin cut . basic principles 1 Occlusive stress maximum distribution in centric relation 2 The occlusive strengths should by the teeth's major axis.3 When the contact is surface to surface, it must be exchanged to another surface point. 4 Once the stability to the centric relation is achieved, it should be kept. The rules to guide the occlusal adjustment selective grinding .
  Arms: Occlusal adjustment
Behavioral: Visual analog scale. — Visual analog scale-Graduation was held on the visual analogue scale in the first and last query to measure discomfort chewing.Graduation was held on the visual analogue scale .in the first and last query to measure discomfort chewing. After graduating dental cleaning was performed, with the purpose of blinding the study, Dental Cleaning.With engine using low speed, brushes, and prophylactic paste is carried out dental cleaning in the teeth of all patient.
  Dental Cleaning.With engine using low speed, brushes, and prophylactic paste is carried out dental cleaning in the teeth of all patient.

SUMMARY:
* The purpose of this study was to evaluate the effects of Neuro Occlusal Rehabilitation (RNO) in patients with peripheral facial palsy (PFP) disease, noting the decrease in symptoms of masticatory dysfunction.
* According to Carvalho (2009) patients with PFP have chronic unilateral masticatory preference. Santos et al. (2009) in the same year noted that these conditions can lead to problems with temporomandibular disorder.
* Hypothesis- known that performing occlusal adjustment in these patients with chronic PFP, ensuring a maximum of dental contacts and a final stop of the masticatory cycle stable, providing a balanced occlusion.
* dental cleaning was performed in two groups for the blind study
* visual analog scale -To assess the quality of the oral functions of these patients, the investigators applied the visual analog scale(VAS) and statistically evaluated the degree of satisfaction regarding the functions of oro facial in relation to mastication and temporomandibular dysfunction.
* gnathostatic models were made in the treatment group in the first and last query.
* occlusal adjustment in treatment group.In the group treated occlusal adjustment was made in the teeth and applied a new (VAS) before and after treatment.

The RNO, is defined as a part of medicine that operates in stomatology occlusal plane as a guide to a harmonious development of the face, chewing facilitating bilateral and alternating. (Planas, 1997). It works through selective grinding on the occlusal platform, providing an increased number of dental contacts.

DETAILED DESCRIPTION:
Purpose: To evaluate the effects of the Neuro-Rehabilitation occlusion in patients with chronic facial palsy by observing the decrease of the symptoms of masticatory dysfunction.

Methods: a selection of sixty-five patients with facial palsy (PFP 65) and idiopathic chronic trauma of the Otorhinolaryngology sector facial nerve disorders at UNIFESP.

Patients were of both genders, aged between 18 and 60. They were analyzed according to the criteria of inclusion and exclusion, resulting in forty-three patients.

However, due to problems inherent in research, a group of fourteen patients were randomized (sub-divided) into two groups: control and treatment.

The visual analog scale was used at the first consultation to patients in the control and treatment group.

All patients underwent a dental cleaning in order to blind the study. Seven patients belonged to the control group for three months per sequence, the VAS was performed in both groups. The control group was later reunited with the treatment group after three months of control period, increasing the number of patients who were examined in extracts, with similar features in a prognostic factor.

* Control group
* First visit- visual analogue scale and dental cleaning - Day 1
* Second visit, after a month, a new visual analog scale. Day-30
* Third-visit -one months after a new visual analogue scale Day 60 patient was a three visits with an interval of one month, performing a repeat procedure.

  * Last visit - Day 90 visual analogue scale
* Treatment group The researchers applied the technique of Rehabilitation and Neuro Occlusal gnathostatic models that were made before and after treatment to count the dental contacts.
* First query - visual analogue scale and dental cleaning, preparation of initial models gnatostaticos and intervention- Day 1
* Second-query-after a month, a new visual analogue and intervention. Day 30
* Third query- -after a month, a new visual analogue and intervention Day 60
* Last query -after a month a new visual analogue scale and making models gnathostatic finals. Day 90 The treatment group had one month to see changes in oral functions, but for estatistic effects was computed only de first andy the last visit the number of the dental contact and the VAS. Day 90 Upon completion of the study patients continued to receive care in the ambulatory clinic of the university, but the attendance for this research was terminated.

ELIGIBILITY:
Inclusion Criteria:

* patients with PFP over six months of treatment
* indentations
* carrier fixed partial dentures and removable drives and/or dental implants
* palsy classified as Grade III according to House and Brackmann scale

Exclusion Criteria:

* patients who already had other diseases in the region of the jaws before facial paralysis
* is toothless from installing, using or not dentures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosana Q Costa, master, Principal Investigator — Federal University of São Paulo; Rosana Q Costa, Investigator, Principal Investigator — Federal University São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahal A, Goffi-Gomez MV. Clinical and electromyographic study of lateral preference in mastication in patients with longstanding peripheral facial paralysis. Int J Orofacial Myology. 2009 Nov;35:19-32. PMID 20572435
- [Background] Martin E. [Neuro-occlusal rehabilitation and selective grinding: results after 1 year]. Orthod Fr. 2000 Jan;71(1):57-60. French. PMID 10838864
- [Background] Planas P. [Equilibrium and neuro-occlusal rehabilitation]. Orthod Fr. 1992;63 Pt 2:435-41. French. PMID 1341730
- [Background] Planas M. [Neuro-occlusal rehabilitation: NOR]. Orthod Fr. 1971;42:333-47. No abstract available. French. PMID 5293022
- [Background] Christensen LV, Radue JT. Lateral preference in mastication: an electromyographic study. J Oral Rehabil. 1985 Sep;12(5):429-34. doi: 10.1111/j.1365-2842.1985.tb01548.x. PMID 3862802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was a selection of sixty-five patients with traumatic and idiopathic palsy of the Otorhinolaryngology UNIFESP, between June 2008-March 2009, according to the criteria of inclusion and exclusion, resultram forty-four, of whom 30 did not participate, resulting in 14.
Pre-assignment Details: Some patients were excluded because they did not agree to be randomized, others could not be present at every visit, or were co-interventions.
Groups:
- Placebo Then Treatment: Participants recived, Dental cleaning and performing the visual analog scale, durant tree visits.
  At first visit was doing Dental cleaning and visual analog scale and after 90 days was doing another visual analog scale.
  Participants who recieved Placebo later recieved Treatment as described for The experimental-Occlusal Adjustment Arm.
- Experimental-Occlusal Adjustment: Participants recived, Dental cleaning, occlusal adjustment, and visual analog scale and gnathostatic models in the first visit.
  After three times, consecutively, one visit a month, the intervention was performed. At the first visit and after 90 days, visual analog scale, and gnathostatic models, were performed.
Period: 01-90
Arm/Group | Placebo Then Treatment | Experimental-Occlusal Adjustment
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: 91-180
Arm/Group | Placebo Then Treatment | Experimental-Occlusal Adjustment
Started | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only on the treatment group was done the brand carbon count models, and gnatostatic models.
Groups:
- Control Group-visual Analog Scale (EVA), Dental Cleaning: Dental cleaning and performing the visual analog scale. At first visit was doing Dental cleaning and visual analog scale and after 90 days was doing another visual analog scale.
- Treatment Group-EVA,Dental Cleaning,Occlusal Adjustment.: Dental cleaning, occlusal adjustment, and visual analog scale and gnathostatic models was doing in the intervention group, at the first visit and after 90 days, visual analog scale, and gnathostatic models.
- Total: Total of all reporting groups
Arm/Group | Control Group-visual Analog Scale (EVA), Dental Cleaning | Treatment Group-EVA,Dental Cleaning,Occlusal Adjustment. | Total
Number analyzed (Participants) | 07 | 07 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — The patient's age affects the prognosis, the sample should be as uniform as possible.
  years | 36.6 (9.8) | 36.4 (9.2) | 36.42 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 1 | 6 | 7
Cause of facial paralysis [Number; unit: participants]
  Traumatic | 4 | 3 | 7
  Idiopatic | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Visual Analog Scale for Pain Was Used to Grade Discomfort in Chewing After the Installation of Facial Paralysis. Level Zero is the Lack of Discomfort and 10 is the Maximum Degree of Discomfort.
Description: It is a scale-shaped ruler, which is associated with faces used to grade the degree of pain for patients, before and after treatments, or just graduating pain and its severity for the patient (Souza, 2002).
  Patients were asked to fill the VAS with the following questions.
  * Do you chew well?
  * How would you classify your chewing at the moment?
  * If you have no trouble chewing, the rating is zero.
  * If you have any discomfort when you chew, your reference level is five.
  * If the discomfort is intense, its reference level is ten. The greater the discomfort, the greater the scale.
Time Frame: Day 1 (Day 91 for Treatment participants first receiving Placebo)
Population: All participants were treated by intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo-VAS, Dental Cleaning: Dental cleaning and performing the visual analog scale. At first visit (day 1) was doing Dental cleaning and visual analog scale.
- Treatment- VAS,Dental Cleaning,Occlusal Adjustment.: Dental cleaning, occlusal adjustment, visual analog scale and gnathostatic models was doing in the intervention group, at the first visit.(day 1). After day 90,the control group passed to treatment group, (day 91)and start the treatment and was done dental cleaning, occlusal adjustment, visual analog scale, and gnatostatic models.
Arm/Group | Placebo-VAS, Dental Cleaning | Treatment- VAS,Dental Cleaning,Occlusal Adjustment.
Number analyzed (Participants) | 07 | 14
units on a scale | 5.6 (1.1) | 6.1 (1.8)
Statistical Analysis 1: Comparison: Placebo-VAS, Dental Cleaning vs Treatment- VAS,Dental Cleaning,Occlusal Adjustment; We assessed the quality of oral functions in the first query to check the status of discomfort before treatment in both groups, using VAS.. Statistical significance was considered for values of p <0.05 and it was used The Minitab statistical software, version 15.1 to obtain the results; Test type: Equivalence — The comparison among the groups, from the results obtained by the Visual Analog Scale (VAS), was done through analysis of variance models (ANOVA) with two factors; p = 0.524, t-test, 1 sided — Statistical significance was considered for values of p <0.05 and it was used The Minitab statistical software, version 15.1 to obtain the results; The comparison between the groups in each study period (initial) was done through the t-test for two independent samples; Mean Difference (Net) = 0.5

2. Primary Outcome: Brand Carbon Count on Gnathostats Models
Description: Only in the treatment group were done gnatostatic models.The models were placed occluding brought with carbon, using the willis compass to keep occluding the posterior base of the model which are aligned with the rear. A model of the teeth was made to measure the occlusion of the teeth (i.e., the amount of contact between the upper and lower mandibles), and used carbon to count the the number of dental contacts, through the brand carbon made on the model, The dental contacts were counted in the models before and after treatment. The models are made in the first and last query.
Time Frame: Day 01 and after 90 days of treatment (Day 180 for Treatment participants first receiving Placebo)
Measure: Mean (Standard Deviation); unit: number of dental contacts
Groups:
- First Query: The dental contacts were evaluated in models and gnathostats demarcated after the points were counted in the models before the treatment.
  The models are made in the first query (day 1, and day 91).The models were placed occluding brought with carbon, using the willis compass to keep occluding the posterior base of the model which are aligned with the rear. A model of the teeth was made to measure the occlusion of the teeth (i.e., the amount of contact between maxilla and mandible) and used carbon marks to count the the number of dental contacts.
- Last Query: The dental contacts were evaluated in gnathostats models and demarcated , the points were counted in the models after treatment. A model of the teeth was made to measure the occlusion of the teeth (i.e., the amount of contact between the upper and lower mandibles), and used carbon to count the the number of dental contacts.
  The models are made on last query,(day 90 to treatment group, and day 180 to controll group turn to be treatment) after four visits on treatment group with one month interval between them.
  The models were placed occluding brought with carbon, using the willis compass to keep occluding the posterior base of the model which are aligned with the rear.
Arm/Group | First Query | Last Query
Number analyzed (Participants) | 14 | 14
number of dental contacts | 9.6 (3.0) | 14.6 (4.4)
Statistical Analysis 1: Comparison: First Query vs Last Query; The brand carbon mark was done on the treatment group in the first and last query; Test type: Equivalence — Only the treatment group was analysed. The dental contacts were evaluated in models and gnathostats demarcated after the points were counted in the models before and after treatment If an increase in the number of dental contacts after occlusal adjustment was detected, in relation of the models. The models are made in the first and last query, after four visits with one month interval between them; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 5, Standard Deviation 3.92

3. Secondary Outcome: Visual Analog Scale
Description: It is a scale-shaped ruler, which is associated with faces used to grade the degree of pain for patients, before and after treatments, or just graduating pain and its severity for the patient (Souza, 2002).
  Patients were asked to fill the VAS with the following questions. Do you chew well? How would you classify your chewing at the moment? If you have no trouble chewing, the rating is zero. If you have any discomfort when you chew, your reference level is five. If the discomfort is intense, its reference level is ten. The greater the discomfort, the greater the scale.
Time Frame: After 90 days of treatment (Day 180 for Treatment participants first receiving Placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo-Vas, Dental Cleaning: Dental cleaning and performing the visual analog scale. At first visit (day 1) was doing Dental cleaning and visual analog scale and after 90 days was doing another visual analog scale.
- Treatment VAS,Dental Cleaning,Occlusal Adjustment.: Dental cleaning, occlusal adjustment, and visual analog scale and gnathostatic models was doing in the intervention group.
  Day 1 and day 90, to treatment group; And day 91 and day 180 to controll group that passed to treatment group.
Arm/Group | Placebo-Vas, Dental Cleaning | Treatment VAS,Dental Cleaning,Occlusal Adjustment.
Number analyzed (Participants) | 07 | 14
units on a scale | 5.4 (1.3) | 3.0 (1.5)
Statistical Analysis 1: Comparison: Placebo-Vas, Dental Cleaning vs Treatment VAS,Dental Cleaning,Occlusal Adjustment; We assessed the quality of oral functions in the last query to check the status of discomfort after ninety days in both groups, control and treatment, using VAS. The statistical significance was considered to p<0.05 values and it was used the Minitab statistics software, 15.1 version, to get the results; Test type: Equivalence — The comparison among the groups, from the results obtained by the Visual Analog Scale (VAS), was done through analysis of variance models (ANOVA) with two factors. The comparison among the groups, in each period of the study (initial and final) was done through t test for two independent samples; p = 0.002, t-test, 2 sided; Mean Difference (Net) = 2.4, Standard Deviation 1.44

4. Other Pre Specified Outcome: Correlation Between the Increase of the Number of Dental Contact Points and the Improvement in the Subjective Evaluation Measured Through the Visual Analogic Scale .
Description: The correlation between the increase of the number of the dental contacts and the VAS evaluation final result from chronic peripheral facial paralysis patients, according to control and treated groups by the neuro occlusal rehabilitation technic.
Time Frame: Day 01 and after 90 days of treatment (Day 180 for Treatment participants first receiving Placebo)
Measure: Number; unit: correlation coefficient
Groups:
- Treatment-VAS Dental Cleaning Occlusal Adjustment: Dental cleanning, occlusal adjustment, and visual analog scale and gnathostatic models was doing in the intervetion group, at the first visit and after 90 days, visual analog scale, and gnathostatic models.
Arm/Group | Treatment-VAS Dental Cleaning Occlusal Adjustment
Number analyzed (Participants) | 14
correlation coefficient | 0.111
Statistical Analysis 1: Comparison: Treatment-VAS Dental Cleaning Occlusal Adjustment; Test type: Other; p = 0.705, t-test, 1 sided

5. Other Pre Specified Outcome: Correlation Between the Increase of the Number of Dental Contact Points and the Improvement in the Subjective Evaluation Measured Through the Visual Analogic Scale Whithout the Outlier.
Description: The correlation between the increase of the number of the dental contacts and VAS evaluation final result from chronic peripheral facial paralysis patients.
  On this measure was excluded one outlier patient whose facial paralysis appeared in her childhood.
  Observing the outlier patient, it was carried out a new scatterplot, ignoring her.
Time Frame: Day 01 and after 90 days of treatment (Day 180 for Treatment participants first receiving Placebo)
Measure: Number; unit: correlation coefficient
Arm/Group | Treatment-VAS Dental Cleaning Occlusal Adjustment
Number analyzed (Participants) | 13
correlation coefficient | 0.638
Statistical Analysis 1: Comparison: Treatment-VAS Dental Cleaning Occlusal Adjustment; Test type: Other; p = 0.01, t-test, 1 sided

ADVERSE EVENTS:
Groups:
- Visual Analog Scale, Dental Cleaning: Dental cleaning and performing the visual analog scale. At first visit was doing Dental cleaning and visual analog scale and after 90 days was doing another visual analog scale.
- Visual Analog Scale,Dental Cleaning,Occlusal Adjustment.: Dental cleaning, occlusal adjustment, and visual analog scale and gnathostatic models was doing in the intervention group, at the first visit.
  After 90 days, visual analog scale, and gnathostatic models, was doing again.
Arm/Group | Visual Analog Scale, Dental Cleaning | Visual Analog Scale,Dental Cleaning,Occlusal Adjustment.
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/14
Other Adverse Events (participants affected / at risk) | 0/7 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No